CLINICAL TRIAL: NCT02794038
Title: Accuracy & Usability Study for Soberlink Cellular Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soberlink Healthcare LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: ACUSPROT 2016-001
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soberlink Cellular Device (Active Comparator): BAC reading with Soberlink Cellular Device
  Interventions: Device: BACtrack S80 Pro
- BACtrack S80 Pro (Active Comparator): BAC reading with BACtrack S80 Pro
  Interventions: Device: Soberlink Cellular Device

INTERVENTIONS:
Device: Soberlink Cellular Device — BAC breath analyzer
  Arms: BACtrack S80 Pro
Device: BACtrack S80 Pro — BAC breath analyzer
  Arms: Soberlink Cellular Device

SUMMARY:
This study scope is to validate the accuracy and usability of the Soberlink Cellular Device in comparison to a predicate device, BACtrack S80 Pro.

DETAILED DESCRIPTION:
The purpose of this accuracy and usability study is to validate the performance of Soberlink Cellular Device in the hands of the intended (lay) users - untrained study participants who have consumed alcohol and use the Soberlink Cellular Device to measure their blood alcohol content (BAC) in comparison to a predicate device.

The purpose of this document is to define how the human factors environment impacts the actual user interface design as well as how usability engineering evaluates user interface via usability objectives and usability tests. This accuracy and usability study will be performed on Soberlink Cellular Device in order to comply with FDA's Draft Guidance for Industry and Food and Drug Administration Staff, titled: Applying Human Factors and Usability Engineering to Optimize Medical Device Design, IEC 60601-1-6 (collateral standard for usability engineering of medical electrical equipment), and IEC 62366 (application of usability engineering to medical devices).

ELIGIBILITY:
Inclusion Criteria:

* Subject willing to sign an informed consent
* Male or female subject between the ages of 21-99 years old
* Untrained subject in the use of an Alcohol Breathalyzer
* Subject willing to consume two alcoholic drinks
* Subjects willing to use two Alcohol Breathalyzers
* Subject willing to complete a Questionnaire

Exclusion Criteria:

* Subject with previous Alcohol Breathalyzer experience
* Subject currently in substance use rehabilitation or post rehabilitation, or unauthorized to consume alcohol for any other reason
* Subject with lung disease, or is physically unable to provide a deep lung exhalation for 4 seconds
* Subject unwilling to drink two alcoholic drinks
* Subject unwilling to complete a questionnaire
* Subject that is non-English speaking
* Subject that is a child, adolescent, or cognitively impaired.
* Subject that is a pregnant and/or breastfeeding woman

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Validate the accuracy of the Soberlink Cellular Device in comparison to a predicate device, BACtrack S80 Pro and assessed by linear regression. | Day 1
  Performance validation will occur by evaluating the accuracy of the Soberlink Cellular device in the hand of intended users - untrained study participants who have consumed alcohol and use the device to measure their blood alcohol content (BAC). 40 adults will be recruited who have recently consumed alcohol. The only assistance to be provided is the labeling. No additional coaching, either written or verbal, will be provided to study participants. Participants should obtain a BAC reading with the Soberlink Cellular device, and a second BAC reading with a comparator device. The second measurement will be taken within 5 minutes of the first. A linear regression line for the comparison between results of the Soberlink Cellular device and a comparator will be made.

SECONDARY OUTCOMES:
Validate the usability of the Soberlink Cellular Device in comparison to a predicate device, BACtrack S80 Pro and assessed by Questionnaire. | Day 1
  Performance validation will occur by evaluating the usability of the Soberlink Cellular device in the hand of intended users - untrained study participants who have consumed alcohol and used the device to measure their blood alcohol content (BAC). 40 adults who have recently consumed alcohol will be asked to evaluate the Soberlink Cellular device. The only assistance provided is the labeling. No additional coaching, either written or verbal, will be provided to study participants. Participants should obtain a BAC reading with the Soberlink Cellular device, and a second BAC reading with a comparator device. The second measurement should be taken within 5 minutes of the first. Following the second measurement a questionnaire will be administered to study participants to evaluate the ease of use of the Soberlink Cellular device.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Hanrahan, PhD, Principal Investigator — Private Practice

IPD SHARING:
Plan to Share IPD: Yes
Participant will be aware of their own BAC result as the result is displayed on the LED screen of the device